CLINICAL TRIAL: NCT02003599
Title: Laser InGaAlP (660Nm) to Prevent Radiodermatitis in Breast Cancer Patients Submitted to Radiation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Vale do Sapucai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MPMarina
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2015-05

CONDITIONS: Radiotherapy; Adverse Effect, Dermatitis or Eczema; Breast Neoplasms
Keywords: Radiodermatitis; Breast neoplasms; Laser Therapy, Low- Level
MeSH Terms: conditions — Dermatitis; Eczema; Breast Neoplasms; Radiodermatitis | interventions — Laser Therapy; Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): In the control group, 26 patients will be submitted to a laser, but the laser will be disabled without affecting its apparent function , five days a week before radiotherapy .
  Both arm will use institutional skin care protocol.
  Interventions: Device: Placebo
- Laser therapy (Experimental): In the intervention group, 26 patients will be submitted a laser therapy .The low level laser therapy used in this trial will be Photon Lase III (DMC, approved by ANVISA for medicinal purposes). This InGaAIP laser emits a pulsed 660 nanometer beam with an average output of 80 milliwatts and the average energy density delivered to the breast will be 3 J/cm2. It will be administrated five days a week before radiotherapy.
  Both arm will use institutional skin care protocol.
  Interventions: Device: Laser therapy

INTERVENTIONS:
Device: Laser therapy — The low level laser therapy used in this trial will be Photon Lase III (DMC, approved by ANVISA for medicinal purposes). This InGaAIP laser emits a pulsed 660 nanometer beam with an average output of 80 milliwatts and the average energy density delivered to the breast will be 3 J/cm2.
  Other Names: Low-Level Laser Therapy; Low Level Laser Therapy; LLLT
  Arms: Laser therapy
Device: Placebo — In the control group, 26 patients will be submitted to a laser, but the laser will be disabled without affecting its apparent function , five days a week before radiotherapy .
  Other Names: Placebo Treatment
  Arms: Placebo

SUMMARY:
Breast neoplasm is the second most common type in the world. Radiation therapy is a key component in the treatment of breast cancer. Acute skin reaction is one of the most common side effects of radiation therapy. Several studies were performed for prophylaxis of this adverse event, however, until this moment there is no consensus for clinical practice . Second meta-analysis , the ideal candidate for the radiodermatitis prevention would be an agent capable of repairing damage to DNA or agents that promote cell proliferation . The low power laser promotes tissue repair ( reduces inflammatory phase and induces collagen synthesis ) . Its use in the treatment of adverse events of cancer treatment is well established in two situations : in the prophylaxis and treatment of mucositis and in the treatment of lymphedema . The purpose of this study is to use the low power laser in patients with breast cancer undergoing radiotherapy treatment to evaluate the effects of Laser InGaAIP 660Nm in preventing radiodermatitis.

DETAILED DESCRIPTION:
This study will be a prospective double- blind trial. Patients with breast cancer with stages I-III undergoing to radiotherapy will be included. The participants will be allocated into an intervention group (laser therapy in 26 patients) or a control group ( in 26 patients the laser will be disabled without affecting its apparent function) , five days a week before radiotherapy . The low level laser therapy used in this trial will be Photon Lase III (DMC, approved by ANVISA for medicinal purposes). This InGaAIP laser emits a pulsed 660 nanometer beam with an average output of 80 milliwatts and the average energy density delivered to the breast will be 3 J/cm2. Skin reactions will be graded weekly by a nurse, by a radiotherapist and by an oncologist using the common toxicity criteria (CTC -developed by the National Cancer Institute ) and Acute Radiation Morbidity Scoring Criteria (developed by Radiation Therapy Oncology Group). The patients will answer the modified visual analogue scale for pain (patient self-evaluation).

ELIGIBILITY:
Inclusion Criteria:

1. Age at least 18 years, female gender only.
2. Patients with histological diagnosis of breast cancer (invasive ductal carcinoma, invasive lobular and other types), stages I-III
3. Patients who underwent breast-conserving surgery or mastectomy without breast reconstruction
4. Patients undergoing to adjuvant radiotherapy with conventional dose according to Barretos Cancer's Hospital protocol
5. Patients in the radiotherapy planning , presenting :

   * In the central court : " Hot Spot " ( ICRU ) ≤ 107 %
   * At full volume : " Hot Spot " ( ICRU ) ≤ 110 %

Exclusion Criteria:

* Patients undergoing mastectomy with immediate breast reconstruction
* Patients without histological diagnosis of breast cancer
* Patients with indication for radiotherapy without conventional dose
* Patient with indication for treatment in supraclavicular fossa
* Patients suffering from collagen
* Patients who do not meet the criteria for planning radiotherapy

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-05; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Evaluate the effects of Laser InGaAIP 660Nm in preventing radiodermatitis in women submitted to adjuvant radiotherapy. | 3 months
  Skin reactions will be graded weekly by a nurse, by a radiotherapist and by an oncologist using the common toxicity criteria (CTC -developed by the National Cancer Institute ) and Acute Radiation Morbidity Scoring Criteria (developed by Radiation Therapy Oncology Group).

SECONDARY OUTCOMES:
Evaluate the effects of Laser InGaAIP 660Nm in decreased pain secondary to radiodermatitis | 3 months
  Pain will be graded weekly by the patient.The patients will answer the modified visual analogue scale for pain (patient self-evaluation) (FERRAZ, 1990).

CONTACTS AND LOCATIONS:
Overall Officials: Marina M Costa, MD, Principal Investigator — Universidade do Vale do Sapucaí
Locations (1):
- Hospital do Cancer de Barretos, Barretos, São Paulo, Brazil

REFERENCES:
- [Derived] Costa MM, Silva SB, Quinto AL, Pasquinelli PF, de Queiroz dos Santos V, de Cassia Santos G, Veiga DF. Phototherapy 660 nm for the prevention of radiodermatitis in breast cancer patients receiving radiation therapy: study protocol for a randomized controlled trial. Trials. 2014 Aug 20;15:330. doi: 10.1186/1745-6215-15-330. PMID 25141962